CLINICAL TRIAL: NCT01269073
Title: Comparison Of The Berlin Questionnaire To The Portland Sleep Quiz In Identification Of Patients At Risk For Obstructive Sleep Apnea
Brief Title: Comparison Of The Berlin Questionnaire To The Portland Sleep Quiz
Status: Withdrawn | Type: Observational
Sponsor: Akram Khan (Other)
Responsible Party: Sponsor-Investigator, Akram Khan, Akram Khan, MD, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Other Study IDs: IRB00005628
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Sleep Apnea
Keywords: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This trial is enrolling patients who are already being seen at OHSU sleep disorder center or have been referred for clinical reasons by their physician to the OHSU sleep disorder center and are going to have a sleep study that would be paid for by their insurance company for clinical reasons.

The purpose of this study is to determine whether the Portland sleep apnea quiz has a higher specificity and negative predictive value then the Berlin Sleep Questionnaire in a patient population with a high predisposition to sleep apnea presenting to a sleep center.

DETAILED DESCRIPTION:
This trial is enrolling patients who are already being seen at OHSU sleep disorder center or have been referred for clinical reasons by their physician to the OHSU sleep disorder center and are going to have a sleep study that would be paid for by their insurance company for clinical reasons.

400 consecutive adult subjects who have been referred by their doctor to the sleep disorder center and are undergoing a diagnostic sleep study at the OHSU sleep disorders center will be requested to fill out both a Berlin questionnaire and Portland sleep quiz on the night of the initial diagnostic polysomnography. The questionnaires will be collected and scored in a confidential manner. The predictive value of the questionnaires will be compared with the results of overnight polysomnography (Apnea Hypopnea Index).

ELIGIBILITY:
Inclusion Criteria:

* Adults more than 18 years old

Exclusion Criteria:

* Subjects Unwilling to Complete the Questionnaire

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults presenting to a sleep center
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of 2 questionnaires | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States